CLINICAL TRIAL: NCT07155265
Title: ClinicalTrials.Gov PRS Field-by-Field Checklist & Results Module Templates - REMIMID-ICU
Brief Title: REMIMID-ICU: Remimazolam vs Midazolam for Deep Sedation in Hemodynamically Unstable, Mechanically Ventilated Adults
Acronym: REMIMID-ICU
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yancheng First People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Yiqiu, graduate student, Yancheng First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YCSYY-【2025】-(J-050)
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Mechanical Ventilation; Shock
MeSH Terms: conditions — Critical Illness; Shock | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A - Remimazolam (Experimental): Continuous IV infusion; start 0.10 mg/kg/h and titrate every 15-30 minutes in 0.025-0.05 mg/kg/h steps to target RASS -3 to -5 (allowable range -2 to -5 for clinical safety). Maximum typical rate 0.20 mg/kg/h; temporary higher rates permitted per protocol for breakthrough agitation.
  Interventions: Drug: Remimazolam Besylate
- Arm B - Midazolam (Experimental): Continuous IV infusion; start 0.04 mg/kg/h and titrate every 15-30 minutes in 0.01-0.03 mg/kg/h steps to target RASS -3 to -5 (allowable range -2 to -5). Maximum typical rate 0.20 mg/kg/h per protocol.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam Besylate — Continuous IV infusion; start 0.10 mg/kg/h and titrate every 15-30 minutes in 0.025-0.05 mg/kg/h steps to target RASS -3 to -5 (allowable range -2 to -5 for clinical safety). Maximum typical rate 0.20 mg/kg/h; temporary higher rates permitted per protocol for breakthrough agitation.
  Arms: Arm A - Remimazolam
Drug: Midazolam — Continuous IV infusion; start 0.04 mg/kg/h and titrate every 15-30 minutes in 0.01-0.03 mg/kg/h steps to target RASS -3 to -5 (allowable range -2 to -5). Maximum typical rate 0.20 mg/kg/h per protocol.
  Arms: Arm B - Midazolam

SUMMARY:
This trial evaluates whether remimazolam provides superior sedation quality compared with midazolam in adults receiving invasive mechanical ventilation with ongoing vasopressor support. The primary outcome is the percentage of time within target sedation (RASS -3 to -5) without rescue sedative during the first 48 hours after randomization. Key secondary outcomes include vasopressor exposure (NEE AUC 0-48h), time to awakening, delirium incidence, ventilator-free days, and 28-day mortality.

ELIGIBILITY:
Inclusion

* Age ≥18 years.
* Invasive mechanical ventilation at randomization; anticipated continuous sedation ≥24 hours.
* Hemodynamic instability requiring vasopressor support despite adequate resuscitation: NEE ≥0.10 μg/kg/min for ≥1 hour within 6 hours prior to randomization, or equivalent.
* At least one sign of hypoperfusion (e.g., lactate >2 mmol/L, oliguria, mottled skin, or altered mentation) unless solely due to sedation.

Exclusion

• Known pregnancy; status epilepticus; severe hepatic failure (Child-Pugh C) or on ECMO; refractory hypoxemia requiring prone position at randomization; benzodiazepine hypersensitivity; need for continuous neuromuscular blockade >24h at baseline; moribund not expected to survive 24h; investigator judgement.

Sexes Eligible: All Accepts Healthy Volunteers: No Ages: 18 Years and older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of time within target sedation without rescue | 0-48 hours post-randomization
  Proportion (%) of all valid RASS assessments that are within -3 to -5 with no rescue sedative in the prior 60 minutes, during 0-48h after randomization.

IPD SHARING:
Plan to Share IPD: Yes